CLINICAL TRIAL: NCT05954299
Title: Vincere Biobank Research Protocol
Status: Recruiting | Type: Observational
Sponsor: Vincere Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: VCC-BIOBANK-001
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Cancer; Biobank; Biorepository
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Current blood (plasma, red blood cells), urine, and/or tissue; with the opportunity to collect other biospecimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: Participants and donor samples without disease (ex: non-cancer)
- Disease state or condition: Participants and donor samples with known disease or condition (ex: cancer)

SUMMARY:
The Vincere Biobank aims to make quality biospecimens and associated clinical data available for research studies related to advancing medicine and improving care for patients, including cancer screening, treatment, and care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older; any gender
* Able to donate a blood, urine, tissue, and/or other biospecimen sample
* Able to provide informed consent to participate in the study

Exclusion Criteria:

* Minors, under the age of 18 years
* Individuals who lack the capacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults age 18 years and older of any gender and demographic group, including both healthy participants and those with disease.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Biobank | 10 years
  Collect quality biospecimens with associated clinical data for research studies related to improving medicine and care to the patient, including cancer screening, treatment, and care.

CONTACTS AND LOCATIONS:
Overall Officials: Vershalee Shukla, MD, Principal Investigator — Vincere Cancer Center
Locations (1):
- Vincere Cancer Center, Scottsdale, Arizona, United States